CLINICAL TRIAL: NCT04830644
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Study to Evaluate the Efficacy and Safety of Iguratimod in Patients With Active Primary Sjogren's Syndrome.
Brief Title: A Study to Evaluate the Efficacy and Safety of Iguratimod Compared to Placebo in Patients With Active Primary Sjogren's Syndrome.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM 1910-08-Ⅱ
Record Dates: First submitted 2021-03-28; First posted 2021-04-05 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Primary Sjögren Syndrome
MeSH Terms: interventions — iguratimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Iguratimod 1 (Experimental): orally 25mg twice a day
  Interventions: Drug: Iguratimod
- Iguratimod 2 (Experimental): orally 20mg twice a day
  Interventions: Drug: Iguratimod
- Iguratimod 3 (Experimental): orally 10mg twice a day
  Interventions: Drug: Iguratimod
- Placebo (Placebo Comparator): orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iguratimod — Iguratimod orally twice a day
  Arms: Iguratimod 1; Iguratimod 2; Iguratimod 3
Drug: Placebo — Placebo orally twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of iguratimod compared to placebo in patients with active primary Sjogren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* meet the 2016 American College of Rheumatology (ACR) / European League Against Rheumatism Classification Criteria for Sjogren's Syndrome (EULAR SS)
* ESSDAI score ≥6
* IgG >16 g/L
* Positive anti-SS-A/Ro antibody at screening

Exclusion Criteria:

* Pregnancy or breast feeding
* Secondary Sjogren's syndrome
* severe renal or haematological failure, a history of cancer, hepatitis B or C, human immunodeficiency virus, severe diabetes or any other chronic disease or evidence of infection
* Prior administration of any of the following:

  1. Rituximab in the past 12 months prior to randomization;
  2. Cyclophosphamide, mycophenolate mofetil, methotrexate, leflunomide and iguratimod in the past 12 weeks prior to randomization;
  3. Azathioprine, cyclosporin, tacrolimus, sirolimus, sulfasalazine in the past 4 weeks prior to randomization;
  4. live vaccine in the past 12 weeks prior to randomization
* Corticosteroids: > 10 mg/day oral prednisone (or equivalent); Any change or initiation of new dose within 4 weeks prior to randomization; Intramuscular, subcutaneous, intravenous, or intra-articular corticosteroids within 4 weeks prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) | Week 12
  The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) total score is calculated as the sum of scores for activity level for each domain.
  Overall score, which can range from 0 to 123, a higher score indicates more disease activity

SECONDARY OUTCOMES:
Change From Baseline in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | Week 12
  The total score EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) is calculated as the mean of the 3 individual components.
  Total Score Range (0 = Best outcome and 10 = Worst Outcome)
  The scores for the ESSPRI individual components will be used as such reported by the participants and entered in the case report form (CRF), without any further calculations. It consists of 3 questions covering cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain. Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and overall score is calculated as the mean of 3 individual domains.
Change From Baseline in the Unstimulated Salivary Flow | Week 12
  The mean change from baseline in unstimulated whole salivary flow at all measured time points up to Week 12
Change From Baseline in Schirmer's Test | Week 12
  The Mean change from baseline in Schirmer's Test at all measured time points up to Week 12
  The length in millimeters that the strip wets during the 5 minute test period for each eye. Collection is done separately for each eye.
Change From Baseline in the level of immunoglobulin (IgG, IgA, IgM) | Week 12
  The change from baseline in the level of immunoglobulin (IgG, IgA, IgM) at all measured time points up to Week 12
Change From Baseline in the level of rheumatoid factor (RF) | Week 12
  The change from baseline in the level of RF at all measured time points up to Week 12
Change From Baseline in the level of B -cell activation factor (BAFF) | Week 12
  The change from baseline in the level of BAFF at all measured time points up to Week 12
Change From Baseline in the level of T/B/NK cell subsets | Week 12
  The change from baseline in the level of T/B/NK cell subsets at all measured time points up to Week 12
Change From Baseline in the level of erythrocyte sedimentation rate (ESR) | Week 12
  The change from baseline in the level of ESR at all measured time points up to Week 12
Change From Baseline in the level of serum complement (C3 and C4) | Week 12
  The change from baseline in the level of serum complement (C3 and C4) at all measured time points up to Week 12

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - the Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hebei General Hospital, Shijiazhuang, Hebei
  - the Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - the First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospitalof Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - the First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital Affliated to Shandong First Medical University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - the Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Bethune hospital, Taiyuan, Shanxi
  - the Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - the Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Jiaxing University, Jiaxing, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - the First People's Hospital of Wenling, Wenling, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang